CLINICAL TRIAL: NCT05504863
Title: Effect of Iron Supplementation During Pregnancy on Neurodevelopmental Status of Babies
Brief Title: RAPIDIRON Trial Follow-up Study: RAPIDIRON-KIDS Study
Acronym: RAPIDIRON-KIDS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Jawaharlal Nehru Medical College (Other); S. Nijalingappa Medical College (Unknown); Raichur Institute of Medical Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: R-2111-07169
Record Dates: First submitted 2022-07-20; First posted 2022-08-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Iron Deficiency Anemia; Neurodevelopmental Abnormality; Autism Spectrum Disorder
Keywords: Anemia; Iron Deficiency Anemia; Intravenous iron; India; Low birth weight; Pediatrics; Neurodevelopment
MeSH Terms: conditions — Anemia, Iron-Deficiency; Autism Spectrum Disorder; Anemia | interventions — ferric carboxymaltose; iron isomaltoside 1000; ferric derisomaltose; ferric sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RAPIDIRON IV iron intervention arm 1: Maternal participants in this arm were given a single dose of an IV iron formulation - ferric carboxymaltose - during pregnancy as part of their participation in the parent RAPIDIRON Trial. Participants weighing 50kg and over received a single dose having 1000mg of iron, with others receiving a lower dose as determined by a formula used by the manufacturer (20mg iron/kg body weight). This was given between 14 and 17 weeks fetal gestational age.
  Interventions: Drug: Ferric carboxymaltose
- RAPIDIRON IV iron intervention arm 2: Maternal participants in this arm were given a single dose of an IV iron formulation - iron isomaltoside - during pregnancy as part of their participation in the parent RAPIDIRON Trial. Participants weighing 50kg and over received a single dose having 1000mg of iron, with others receiving a lower dose as determined by a formula used by the manufacturer (20mg iron/kg body weight). This was given between 14 and 17 weeks fetal gestational age.
  Interventions: Drug: Iron isomaltoside
- RAPIDIRON active comparator arm: Maternal participants in this arm of the RAPIDIRON Trial were given ferrous sulfate tablets with 60mg elemental iron each and instructed to take two per day (one in the morning and one at night) throughout their pregnancy.
  Interventions: Drug: Ferric Sulfate

INTERVENTIONS:
Drug: Ferric carboxymaltose — As part of the RAPIDIRON Trial, maternal participants randomized to intervention arm 1 were given a single dose of ferric carboxymaltose between 14 and 17 weeks of pregnancy.
  Groups: RAPIDIRON IV iron intervention arm 1
Drug: Iron isomaltoside — As part of the RAPIDIRON Trial, maternal participants randomized to intervention arm 2 were given a single dose of iron isomaltoside between 14 and 17 weeks of pregnancy.
  Other Names: Ferric derisomaltose
  Groups: RAPIDIRON IV iron intervention arm 2
Drug: Ferric Sulfate — As part of the RAPIDIRON Trial, maternal participants randomized to the active comparator arm were given 200 ferrous sulfate tablets immediately after randomization (~12 weeks of pregnancy). Participants were instructed to take two tablets a day, with each tablet containing 60mg elemental iron.
  Other Names: Ferric sulphate
  Groups: RAPIDIRON active comparator arm

SUMMARY:
As a follow-up to the RAPIDIRON Trial (NCT05358509), this study will follow the previously randomized mothers as well as their offspring after birth to assess neurodevelopmental, hematologic, and health outcomes. The study's overarching goal is to determine if the offspring born to RAPIDIRON Trial mothers in the intravenous iron groups, compared to the oral iron group, will achieve superior neurodevelopment, iron stores, and growth at specific time points during the first three years of life. Differences will be assessed between offspring based on the iron deficiency anemia (IDA) treatment of the mother.

DETAILED DESCRIPTION:
The RAPIDIRON-KIDS Study has two primary hypotheses:

1. Infants born to RAPIDIRON Trial maternal participants from the intravenous (IV) iron arms will have higher hemoglobin and ferritin levels at birth (determined by cord blood) and at 4 months of age compared to infants born to mothers in the oral arm; and
2. Offspring born to RAPIDIRON Trial participants who received IV iron treatment will have higher developmental quotients (DQs) on the cognitive domain of the Bayley Scales of Infant Development (BSID) at 2 years of age compared to offspring born to RAPIDIRON Trial participants given oral iron treatment.

The specific aims of this study are as follows:

* To provide evidence that a single-dose of IV iron (either ferric carboxymaltose or iron isomaltoside, also known as ferric derisomaltose) given to pregnant women in the second trimester during the RAPIDIRON Trial will prove more effective for prevention of neonatal and postnatal iron deficiency in the offspring than the oral iron given to pregnant women per the parent trial protocol
* To assess if the offspring of women in the parent trial IV iron arms have better neurodevelopmental outcomes compared to the offspring of women treated with oral iron; and
* To determine longer-term hematologic effects in previously randomized mothers by obtaining ongoing hematologic indices, documented history of transfusion and hospitalization, and quality of life based on the use of a validated instrument.

This study will recruit pregnant mothers currently participating in the RAPIDIRON Trial, who will be approached to give consent for themselves and their offspring for participation in the RAPIDIRON-KIDS Study. Participation in RAPIDIRON-KIDS will involve assessments at birth, 6 weeks, 4 months, 12 months, 24 months, and 36 months of age. In addition to iron status, anthropometry, and questionnaires relating to child feeding and maternal quality of life, the following neurobehavioral tests will be utilized to assess the offspring at various timepoints: Preferential Looking Test, Ages & Stages Questionnaire 3, Bayley Scales of Infant Development, Behavioral Rating Scale, India Scale for Assessment of Autism, and the Child Behavior Checklist for Ages 1.5-5.

Please see the protocol for additional details.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent of the RAPIDIRON Trial participant for their study inclusion and that of their offspring for the RAPIDIRON-KIDS Study
* Expressed intent of the RAPIDIRON Trial participant to remain in the designated Karnataka research are for delivery and during the follow-up period for the RAPIDIRON-KIDS Study to enable participation in study visits
* For the offspring - live-born singleton infants of Karnataka maternal participants randomized and treated in the RAPIDIRON Trial, if consent is provided by the mother

Exclusion Criteria:

* Unwillingness of maternal participant to provide RAPIDIRON-KIDS Study consent for herself and her offspring

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants of this study are mother-infant dyads consisting of women, residing in Karnataka State (India), who were randomized and treated for iron-deficiency anemia (IDA) during the RAPIDIRON Trial and their newborns.
Sampling Method: Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Offspring hemoglobin | Birth
  Offspring hemoglobin concentration in g/dL
Offspring hemoglobin | 4 months of age
  Offspring hemoglobin concentration in g/dL
Offspring ferritin | Birth
  Offspring serum ferritin concentration in ng/mL
Offspring ferritin | 4 months of age
  Offspring serum ferritin concentration in ng/mL
Cognitive Domain of Bayley Scales of Infant Development (BSID) | 24 months of age
  Developmental quotient (DQ) on the cognitive domain of the Bayley Scales of Infant Development (BSID), conducted at 24 months of age. The Cognitive Domain of the BSID-IV contains 81 items, each item with a minimum score of 0 and a maximum score of 2. A lower score is a bad outcome and a higher score is a good outcome.

SECONDARY OUTCOMES:
Offspring hemoglobin | 12 months of age
  Offspring hemoglobin concentration in g/dL
Offspring ferritin | 12 months of age
  Offspring serum ferritin concentration in ng/mL
Preferential Looking Time | 4 and 12 months of age
  Performance on Preferential Looking Time assessment - scored as the percentage of time spent looking at the novel object during the test phase
Motor and language domains of the Bayley Scales of Infant Development (BSID) | 24 months of age
  Developmental quotient (DQ) on the motor and language domains of the Bayley Scales of Infant Development (BSID), conducted at 24 months of age. The motor domain of the BSID-IV contains 79 items, and the language domain contains 104 items. Minimum score on each item is 0, maximum score is 2. A lower score is a bad outcome and a higher score is a good outcome.
Bayley Scales of Infant Development (BSID) | 36 months of age
  Developmental quotients (DQs) on all domains of the Bayley Scales of Infant Development (BSID), conducted at 36 months of age. There are 5 domains, each many items. Each item has a minimum score of 0 and a maximum score of 2. A lower score is a bad outcome and a higher score is a good outcome.
Behavior Rating Scale | 24 months of age
  Score on the Behavior Rating Scale, as coded from a video recording undergoing the Bayley Scales of Infant Development (BSID). Each child is rated across nine behavioral domains. The minimum score in each domain is 0 and the maximum score is 5, with higher scores indicating more optimal behaviors.
Ages & Stages Questionnaire 3 | 12 months of age
  Accepted and validated screening tool for neurodevelopment. Minimum score of 0, maximum score of 60. Lower score is a bad outcome, higher score is a good outcome.
Child Behavior Checklist for Ages 1.5-5 | 24 and 36 months of age
  A parent-report questionnaire assessing internalizing and externalizing behaviors. Standardized t-scores will result, with a mean of 50 and standard deviation of 10. Higher scores indicate more symptoms (emotional/behavioral) and a worse outcome.
India Scale of Assessment for Autism | 36 months of age
  A standardized screening tool for autism, validated for the Indian population. 40 items are rated from 1 to 5, with a higher score indicating increasing severity.
Offspring weight | 4, 12, 24, and 36 months of age
  Offspring weight measured in kg
Offspring height | 6 weeks, 4, 12, 24, and 36 months of age
  Offspring height measured in cm
Offspring head circumference | Birth, 4, 12, 24, and 36 months of age
  Offspring head circumference measured in cm
Infant and Young Child Feeding Practices | Birth, 6 weeks, 4, 12, and 24 months of age
  A composite questionnaire used to measure feeding practices based upon breastfeeding, dietary diversity, meal frequency, iron supplementation, and iron-fortified foods.
Maternal hemoglobin concentration | 4, 12, and 24 month visits
  Maternal hemoglobin concentration measured in g/dL
Maternal ferritin | 4, 12, and 24 month visits
  Maternal serum ferritin concentration in ng/mL
Maternal well-being/quality of life | 4 and 12 month visits
  Maternal well-being/quality of life, as measured by the World Health Organization Disability Assessment Schedule II (WHODAS-II). Uses 36 items to measure health and disability across six domains of life - cognitive, mobility, self care, relationship, life activities, and participation. Each item is given a score from 0 to 4, and all item scores are summed. Higher scores mean worse outcomes and higher disability status.

OTHER OUTCOMES:
Offspring hospitalization | Birth to 3 years of age
  Incidence of offspring hospitalization
Maternal hospitalization | Birth to 3 years
  Incidence of maternal hospitalization
Maternal transfusions | Birth to 3 years
  Incidence of maternal blood transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Richard Derman, MD, MPH, Principal Investigator — Thomas Jefferson University
Locations (3):
- India (3):
  - S. Nijalingappa Medical College, Bagalkot, Karnataka
  - Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Raichur Institute of Medical Sciences, Rāichūr, Karnataka

REFERENCES:
- [Derived] Derman RJ, Bellad RB, Bellad MB, Bradford-Rogers J, Georgieff MK, Aghai ZH, Thind S, Auerbach M, Boelig R, Leiby BE, Short V, Yogeshkumar S, Charantimath US, Somannavar MS, Mallapur AA, Pol R, Ramadurg U, Sangavi R, Peerapur BV, Banu N, Patil PS, Patil AP, Roy S, Vastrad P, Wallace D, Shah H, Goudar SS. RAPIDIRON Trial follow-up study - the RAPIDIRON-KIDS Study: protocol of a prospective observational follow-up study. Trials. 2023 Dec 20;24(1):818. doi: 10.1186/s13063-023-07740-z. PMID 38124098

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT05504863/Prot_SAP_000.pdf